CLINICAL TRIAL: NCT02959151
Title: A Single-arm Pilot Clinical Study of Chimeric Antigen Receptor T Cells Combined With Interventional Therapy in Advanced Liver Malignancy
Brief Title: A Study of Chimeric Antigen Receptor T Cells Combined With Interventional Therapy in Advanced Liver Malignancy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai GeneChem Co., Ltd. (Industry)
Collaborators: Shanghai Cancer Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAR-T for liver cancer
Record Dates: First submitted 2016-11-06; First posted 2016-11-08 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Carcinoma, Hepatocellular; Pancreatic Cancer Metastatic; Colorectal Cancer Metastatic
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CAR-T for liver cancer (Experimental): A single dose of CART cells will be administered by vascular interventional therapy or by intra-tumor injection with a dose of （1.25~4）×107 CAR positive T cells/cm3 tumor bulk. The volume of cell products and the time of cell perfusion process lasted would depend on the ways of cell perfused. And an interventional radiologist would operate the cell infusion.
  Interventions: Drug: CAR-T cell

INTERVENTIONS:
Drug: CAR-T cell — CAR-T cells are generated by T cells from the patients or a suitable donor transfected by CAR-lentivirus vectors. There are three options for CAR-targets: GPC3 for hepatocellular carcinoma;mesothelin for pancreatic cancer metastatic; CEA for colorectal cancer metastatic.
  Other Names: chimeric antigen receptor T cells

SUMMARY:
The purpose of this study is to collect the date on the safety and potential effectiveness of CART cells combined with interventional therapy in patients with advanced liver malignancy.

DETAILED DESCRIPTION:
Designer T cells are prepared by PBMC which from patients or suitable donator by leukapheresis, and then activated and re-engineered to express chimeric antigen receptors (CARs). There are three options for CAR-targets: GPC3 for hepatocellular carcinoma; mesothelin for pancreatic cancer metastatic; CEA for colorectal cancer metastatic. Cells are expanded in culture and returned to the participant by vascular interventional therapy or by intra-tumor injection at the dose of （1.25~4）×107 CAR positive T cells/cm3 tumor bulk. The volume of cell products and the time of cell perfusion process lasted would depend on the ways of cell perfused.

ELIGIBILITY:
Inclusion Criteria:

* tumor histological examination confirmed as GPC3/ mesothelin/CEA positive expression;
* persistent cancer after at least one prior standard of care chemotherapy, has no willing for surgery or cannot be suitable for surgery patients
* life expectancy greater than 6 months
* satisfactory organ and bone marrow function as defined by the following: (1) creatinine <1.5mg/dl; (2) cardiac ejection fraction of >55%; (3) hemoglobin>9g/dl, bilirubin 2.0×the institution normal upper limit
* without bleeding disorder or coagulation disorders
* Don't allergy to Radiocontrast agent
* birth control
* Adequate venous access for apheresis, and no other contraindications for leukapheresis
* Voluntary informed consent is given

Exclusion Criteria:

* Pregnant or lactating women
* Concurrent use of systemic steroids. Recent or current use of inhaled steroids is not exclusionary
* patients in the situation of: (1) 30 days before apheresis is still in the period of other antitumor drug observation; (2) patient dont recuperate from earlier acute adverse influence brought by any treatments accepted before
* Four weeks before recruit accepted radiation therapy
* Previously treatment with any gene therapy products
* Feasibility assessment during screening demonstrates<30% transduction of target lymphocytes, or insufficient expansion (<5-fold) in response to CD3/CD28 costimulation
* Any serious, uncontrolled diseases (including, but not limit to, unstable angina pectoris, congestive heart failure, grade III or IV cardiac disease, serious arrhythmia, liver and kidney disorders or metabolic diseases, CNS diseases)
* Patient with severe acute hypersensitive reaction
* Taking part in other clinical trials
* Study leader considers not suitable for this tiral

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-07; Primary Completion 2018-01 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Number of patients with adverse event | 6 weeks
  adverse event is evaluated with CTCAE, version 4.0

SECONDARY OUTCOMES:
Number of patients with tumor response | 8 weeks
  summarize tumor response by overall response rates
Detection of transferred T cells in the circulation using quantitative -PCR | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wentao Li, doctor, Principal Investigator — Fudan University
Locations (1):
- Shanghai Tumor Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided